CLINICAL TRIAL: NCT04568798
Title: Efficacy of Sana Treatment in Fibromyalgia: A Blinded Randomized Controlled Trial
Brief Title: Efficacy of Sana Treatment in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Health (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00105695
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Parallel 2-arm study in which patients will be randomly assigned to either active treatment or Sham control arms.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sana Device (Active Comparator): The Sana Device is an externally worn mask that physically contacts the skin of the face. The Sana Device delivers Audio Visual Stimulation (AVS) in the form of coordinated pulses of light (through closed eyelids) and sound at various frequencies.
  Interventions: Device: Sana Sham Device
- Sana Sham Device (Sham Comparator): The sham treatment device is designed to copy the look and feel of the Sana therapy to a degree that it would be indistinguishable from the true treatment. The sham treatment delivers a series of Audio-Visual Stimulation (AVS) in the form of pulses of light (through closed eyelids) and sound, but that offer no therapeutic effect.
  Interventions: Device: Sana Sham Device

INTERVENTIONS:
Device: Sana Sham Device — Externally worn mask that physically contacts the skin of the face. The Sana Device delivers Audio Visual Stimulation (AVS) in the form of coordinated pulses of light (through closed eyelids) and sound at various frequencies.

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of an experimental device called the Sana Pain Reliever Device (Sana Device) on treating pain due to fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Willing to and capable of providing written informed consent prior to the conduct of any study-related procedures.
* Male or female, 18 to 65 years of age, inclusive.
* Clinical diagnosis of Fibromyalgia given a minimum of 8 weeks prior to Screening.
* Patient must have an average pain severity score of ≥40 and <90 on the 100-point VAS for the last 72 hours prior to Screening.
* Any analgesic therapy must be at approximately stable levels for at least 14 days prior to enrollment and remain steady throughout the study.
* Willing and able to comply with the study requirements, complete study assessments, and participate at scheduled times for the duration of the Treatment Phase.
* Able to understand, speak and read English sufficient for the completion of study assessments.

Exclusion Criteria:

* Pregnant or lactating females as self-reported.
* History or presence of photo-sensitive epilepsy or other photo-sensitive conditions.
* History or presence of condition(s) that may affect balance, such as seizure disorders or vertigo.
* Diagnosis of cancer or active cancer treatment occurring within the last year.
* Surgery or trauma requiring rehabilitation within the last 12 weeks.
* Vision impairments that affect perception of light, color, or brightness in one or both eyes, and differences in visual perception between eyes, at the discretion of the investigator.
* Deafness in one or both ears, perceived differences in hearing between ears, or tinnitus, at the discretion of the investigator.
* Current ear or eye infection, untreated allergies, or acute illness that may affect eyes or hearing (e.g., due to congestion).
* Presence of inflammation or broken skin around the eyes in the area of the mask.
* Presence of narcolepsy or untreated sleep apnea or requiring treatment for sleep apnea such that use of device at bedtime will be interrupted, at discretion of the investigator.
* Participation in any other clinical study in which medication(s) are being delivered or have used an investigational drug or device within the last 30 days.
* Any pending legal action that could prohibit participation or compliance in the study.
* Recent history of or current evidence of suicidal ideation or active suicidal behavior, based on medical history, at the discretion of the investigator.
* Significant medical conditions or other circumstances which, in the opinion of the investigator, would preclude compliance with the protocol, adequate cooperation in the study or obtaining informed consent, or may prevent the patient from safely participating in study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Change in quality of life as measured by the Revised Fibromyalgia Impact Questionnaire (FIQR). | Screening, Baseline, Days 14, 28, 56, 112 and 196.
  Scores are measured on a 100 point scale (0-100) with the lower score (0) indicating no difficulty and the higher score indicating very difficult (100).
  Extreme Fibromyalgia (FM): 75-100, Severe FM: 60-74, Moderate FM: 43-59, Mild FM: 0-42
Change in health system utilization. | Days 28 and 196.
  Utilization is self reported via a Health Care Utilization survey.

SECONDARY OUTCOMES:
Change in anxiety as measured by the Generalized Anxiety Disorder 7 (GAD-7). | Screening, Baseline, Days 14, 28, 56, 112 and 196.
  Seven items are rated from 0 - 3 with a lower score indicating less anxiety and a higher score indicated more anxiety.
Change in depression as measured by the Patient Health Questionnaire 8 (PHQ-8). | Screening, Baseline, Days 14, 28, 56, 112 and 196.
  Eight items are rated from 0 - 3 with a lower score indicating less depression and a higher score indicated more depression.
Change in sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI). | Screening, Baseline, Days 14, 28, 56, 112 and 196.
  Seven component scores are derived from 0 -3. A lower score indicates better sleep quality and a higher score worse sleep quality.
Change in pain as measured by the Brief Pain Inventory (BPI). | Screening, Baseline, Days 14, 28, 56, 112 and 196.
  Scores are measured on a 10 point scale with the lower score indicating less interference due to pain and the higher score indicating complete interference.
Change in pain as measured by the Pain Visual Analog Scale (P-VAS). | Daily (Day 0 - 196)
  Scores are measured on a 100mm VAS. The lower number indicates less pain and the higher number more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kollins, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No